CLINICAL TRIAL: NCT03730428
Title: Drug-related Pneumonitis During mTOR Inhibitor Therapy in Patients With Metastatic Breast Cancer: A Radiographic Patternbased Approach
Brief Title: Everolimus Related Pneumonitis in MBC
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-5
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Everolimus; Pneumonitis
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pneumonitis group: Patients who developed drug-related pneumonitis after treated with everolims
- non-pneumonitis group: Patients who didn't develop drug-related pneumonitis after treated with everolims

SUMMARY:
To study the drug-related pneumonitis during mTOR inhibitor therapy in patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal woman (or premenopausal women treated with LHRHa) diagnosed with HR+，HER2- metastatic breast cancer
2. Treated with everolimus for at least one month in metastatic setting
3. With baseline and at least one follow-up chest CT during everolimus therapy.
4. Complete medical history

Exclusion Criteria:

1. Incomplete medical history
2. Radiographic imaging unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
radiographic pattern | 2 months
  Quantitive measure of lung CT
PFS | 2 months
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided